CLINICAL TRIAL: NCT01388920
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Two Doses of Tesamorelin in Stable Ambulatory COPD Subjects With Muscle Wasting
Brief Title: Efficacy and Safety Study of Tesamorelin in Chronic Obstructive Pulmonary Disease (COPD) Subjects With Muscle Wasting
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on a non-safety related corporate decision.
Sponsor: Theratechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TH9507-CTR-1025
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Muscle wasting
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tesamorelin 2 mg (Experimental): Tesamorelin 2 mg/day
  Interventions: Drug: Tesamorelin
- Tesamorelin 3 mg (Experimental): Tesamorelin 3 mg/day
  Interventions: Drug: Tesamorelin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tesamorelin
  Arms: Tesamorelin 2 mg; Tesamorelin 3 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
A significant proportion of COPD subjects experience muscle wasting, which has been associated with increased morbidity, impaired physical functioning, and a poor quality of life.

Muscle wasting is associated with reduced muscle strength in COPD subjects. In particular, weakness of peripheral muscles has been reported to play an important role in the reduced functional capacity and impaired exercise performance.

The primary objective of this study is to investigate the effect of tesamorelin, in conjunction with exercise training, on lean body mass measured by dual energy x-ray absorptiometry (DXA) scan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 40-75 years (y) inclusive
* Documented diagnosis of moderate to very severe COPD (GOLD stage 2, 3, or 4)
* Stable COPD (i.e., no exacerbation) for at least 6 weeks prior to screening
* Able to participate in a supervised exercise training program
* Evidence of muscle wasting

Exclusion Criteria

* Participation in a pulmonary rehabilitation program or in any supervised exercise program during the 4 months prior to screening
* More than 4 exacerbations in the year prior to screening
* Life-threatening exacerbation in the year prior to screening
* Requirement for long-term oxygen therapy (> 12 hours of oxygen per day)
* Critical illness or co-morbid conditions that may interfere with study conduct or endpoint measurements
* Use of agents known to increase lean body mass within 3 months prior to screening
* Hypopituitarism, history of pituitary tumor/surgery, head irradiation, or severe head trauma

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Casaburi, PhD, MD, Principal Investigator — University of California, Los Angeles

RESULTS

PARTICIPANT FLOW:
Groups:
- Tesamorelin 2 mg: Tesamorelin 2 mg/day for 6 months
- Tesamorelin 3 mg: Tesamorelin 3 mg/day for 6 months
- Placebo: Placebo for 6 monts
Period: Overall Study
Arm/Group | Tesamorelin 2 mg | Tesamorelin 3 mg | Placebo
Started | 1 | 1 | 0
Completed | 1 | 1 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo for 6 months
- Total: Total of all reporting groups
Arm/Group | Tesamorelin 2 mg | Tesamorelin 3 mg | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (0) | 51 (0) |  | 55 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 |  | 1
  Male | 1 | 0 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lean Body Mass at 6 Months
Description: The primary objective of the study was to evaluate the effect of tesamorelin on lean body mass by Dual-energy X-ray absorptiometry (DXA) scan
Time Frame: 6 months
Population: The primary objective of the study was the change in lean body mass between baseline and Month 6. However, the study was halted approximately 1 month after patient enrollment.
Arm/Group | Tesamorelin 2 mg | Tesamorelin 3 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Exercise Capacity at 6 Months
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Peripheral Muscle Strength at 6 Months
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Patient-reported Outcomes at 6 Months
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Adverse Events
Description: Number and percentage of subjects with adverse events
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: COPD Exacerbations
Description: Frequency and severity of COPD exacerbations
Time Frame: 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Plasma Glucose
Description: Changes from baseline in fasting blood glucose
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Tesamorelin 2 mg | Tesamorelin 3 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No